CLINICAL TRIAL: NCT06547255
Title: Exparel Versus Bupivacaine in Post-operative Pain Control Following Bilateral Third Molar Extractions: A Single-blind Randomized Clinical Trial
Brief Title: Exparel Versus Bupivacaine in Post-operative Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Faisal Quereshy, professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20221478
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Liposomal Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard bupivicaine (Active Comparator): patient receive mandibular and maxillary infiltrations with 3mL of standard 3mL standard bupivacaine.
  Interventions: Drug: Bupivacaine liposome injectable suspension
- liposomal bupivacaine (Experimental): patient receive mandibular and maxillary infiltrations with 3mL of 1.3% liposomal bupivacaine (Exparel)
  Interventions: Drug: Bupivacaine liposome injectable suspension

INTERVENTIONS:
Drug: Bupivacaine liposome injectable suspension — At the end of the third molar extraction surgical procedure performed under general anesthesia and at least fifteen minutes following the most recent administration of 2% lidocaine with 1:100,000 epinephrine nerve block (routine for this procedure), all patients will receive bilateral infiltrations with 3mL of 1.3% liposomal bupivacaine (Exparel) OR with 3mL of 0.5% bupivacaine with 1:200,000 epinephrine while they are still under general anesthesia.
  Other Names: standard bupivacaine

SUMMARY:
This is a prospective, randomized study to evaluate anaesthetic parameters, postoperative analgesia and oral analgesic consumption comparing exparel (liposomal bupivacaine) vs. standard bupivacaine

DETAILED DESCRIPTION:
The main purpose of this prospective, randomized study was to evaluate anaesthetic parameters, postoperative analgesia and oral analgesic consumption comparing exparel (liposomal bupivacaine) vs. standard bupivacaine. At the end of the third molar extraction surgical procedure and at least fifteen minutes following the most recent administration of 2% lidocaine with 1:100,000 epinephrine (routine for this procedure), patients will, at random, receive mandibular and maxillary infiltrations with 3mL of 1.3% liposomal bupivacaine (Exparel) or with standard 3mL standard bupivacaine. Electronic home questionnaires will be completed by the patient following the procedure for 96 hours to evaluate these clinical parameters

ELIGIBILITY:
Inclusion Criteria:

* Male and nonpregnant female adults (≥18 years of age) with American Society of Anesthesiologists physical status classification 1, 2, or 3 who were scheduled to undergo bilateral third molar extraction (extraction of all 4 third molars) under local anesthesia and general anesthesia Study participants were required to have full or partial bony impaction of both mandibular third molars.

Exclusion Criteria:

* history of allergy or contraindication to amide-type local anesthetics, epinephrine, or opioids a history of any disease or condition or recent use of any drug that, in the opinion of the investigator, might increase the risk of surgery or interfere with study evaluations any use of long-acting opioids, nonsteroidal anti-inflammatory drugs, aspirin, or acetaminophen within 3 days before screening or use of opioids within 24 hours of screening Patient that is pregnant or suspected to be pregnant Adults that cannot speak English, adults that are unable to consent on their own, or persons that are listed as vulnerable individuals will not be part of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
post operative pain | 96 hours post-operatively
  At home questionnaire with a numerical scale (0 - 10), to be completed each morning and evening for four days post-operative
Adverse effects | 96 hours post-operatively
  At home questionnaire including the presence or absence of any abnormal sensations, change in taste, nausea, constipation, fever, diaphoresis, vomiting, light-headedness, palpitations, or headache.
NSAID/Acetaminophen use | 96 hours post-operatively
  Ibuprofen 600mg [Advil], Tylenol) Use
Norco 5/325 (Hydrocone-Acetaminophen) Use | 96 hours post-operatively
  At home questionnaire including the dosage, time, quantity and reason for use

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Quereshy, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No